CLINICAL TRIAL: NCT01492660
Title: Comparison of Visibility of Echogenic and Standard Non-echogenic Block Needles During Ultrasound Guided Sciatic Blocks. A Randomized Prospective Study
Brief Title: Echogenic Versus Stimulating Needle and Catheter for Sciatic Blocks
Acronym: Echostim1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Sugantha Ganapathy, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-11-495; 17757 (Other: REB)
Record Dates: First submitted 2011-10-11; First posted 2011-12-15 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2012-01

CONDITIONS: Osteoarthritis Knee; Postoperative Pain
Keywords: Ultrasonography; nerve block; catheters; needle; anesthesia
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Catheters

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Echogenic needle and catheter (Experimental): The echogenic needle will be positioned using ultrasonography and neurostimulation with an end point of plantar or dorsiflexion with 0.6mA of current strength. The catheter will be inserted using ultrasonography alone. 20 Ml of 2% mepivacaine will be inserted using the catheter. The distribution of drug will be evaluated using short axis and long axis views. Sensory motor block evaluation every 5 minutes for 30 minutes. Duration of block procedure, number of passes and success will be evaluated
  Interventions: Device: echogenic needle and catheter
- Neurostimulation (Active Comparator): The non echogenic needle will be positioned using ultrasonography and neurostimulation with plantar or dorsiflexion as the end point with 0.6mA current.The catheter will be positioned using neurostimulation with plantar or dorsiflexion with 0.6-1.5mA current.
  Interventions: Device: Neurostimulation to position needle and catheter

INTERVENTIONS:
Device: echogenic needle and catheter — Visibility of needle shaft and tip with engraved markers. Ultrasonographic Visibility of catheter tip
  Other Names: Pajunk Stimulong plexus catheter set; Pajunk sonolong sonoset
  Arms: Echogenic needle and catheter
Device: Neurostimulation to position needle and catheter — The non echogenic needle will be positioned using ultrasonography and neurostimulation and the catheter will be positioned using neurostimulation with plantar or dorsiflexion with 0.6-1.5mA current. 20mL of 2% mepivacaine will be injected via the catheter. Sensory motor block will be evaluated every 5 minutes for 30 mins
  Other Names: Pajunk Stimulaong Plexus catheter set
  Arms: Neurostimulation

SUMMARY:
Patients scheduled for total knee replacements and suitable for sciatic nerve block will be randomized to one of 2 groups.

Group 1 will have the nerve block performed using a standard Pajunk block needle under ultrasound guidance and with electrical nerve stimulation (ENS), and have catheter placement also guided by electrical nerve stimulation. Group 2 will have the block performed using a Sonoplex echogenic block needle and have an echogenic catheter sited, all under ultrasound (US) guidance. Group 2 will have needle location aided by ENS, but ENS will not be used for catheter location.

An observer blinded to the needle type will assess the quality of needle visualisation on a recording of the US image taken during the procedure, along with adequacy of spread of local anesthetic. The primary outcome will be needle visibility, and secondary outcomes will be block success rate, block performance time, complication rate, number of needle passes per block, and adequacy of spread of local anesthetic.

DETAILED DESCRIPTION:
A total of 70 patients with ASA physical status 1 to 4, scheduled for elective total knee arthroplasty and deemed suitable to receive a sciatic nerve block will be included in the study. They will be randomised to one of two groups prior to the block procedure using a closed envelope system.

Recruitment will take place in the preoperative clinic. All blocks will be performed in the block room using standard monitoring, sterile precautions and titrated intravenous sedation.

Prior to the sciatic nerve block a continuous femoral nerve block will be performed according to standard procedure. Once this is complete the patient will be positioned for the sciatic nerve block.

A preprocedural scan will be done as per standard practice and skin will be infiltrated with 1% lidocaine.

The anaesthetist performing the block will be aware of the study group allocation due to the requirement for physically handling the block needles, and will proceed to position the needle into the required location site to facilitate catheter insertion, with the aid of electrical nerve stimulation via the needle. This will be recorded using the ultrasound machines cineloop facility.

If after 6 passes the operator is unable either to contact the nerve according to the ultrasound image or elicit a twitch response, the procedure will be abandoned and this will be considered a failed block. In this case analgesia will be covered with periarticular infiltration and opioids.

During needle positioning, the observer will record the number of needle redirections required to optimally locate the needle, each redirection being defined as every movement which follows a withdrawal of more than 2cm. The observer will also record the number of skin punctures required and any arterial or venous punctures.

Group E will have the block performed using the echogenic needle, and the echogenic catheter will be placed using ultrasound guidance.

The catheter will be inserted through the needle by a second anesthetist. This process will be continuously recording using the cineloop feature of the ultrasound machine. Once the catheter is deemed to be in an appropriate position, local anaesthetic will be injected by the second anaesthetist while observing the disposition of the local anaesthetic perineurally in short axis. This will be confirmed with a long axis view of the nerve (also recorded).

Group S will have the block performed with a standard needle and catheter, guided by electrical nerve stimulation.

Acceptable muscle twitch response will be plantar- or dorsiflexion, inversion or eversion with an initial nerve current strength of 0.5mA at a frequency of 2Hz. If a satisfactory motor response cannot be elicited, current will be increased in stages to 1.5mA. If a response still cannot be elicited this will be recorded but the catheter will still be used if its position is deemed satisfactory using colour Doppler - a medley of colour adjacent to the nerve with the injection of agitated dextrose 5%. Once the catheter is deemed to be in an appropriate position, local anaesthetic will be injected by the second anaesthetist while observing the disposition of the local anaesthetic perineurally in short axis. This will be confirmed with a long axis view of the nerve (also recorded).

Once the catheter has been sited using the above techniques, a bolus of agitated 5% dextrose will be injected through the catheter and Doppler ultrasound will be used to locate where in the tissues the injected fluid is being deposited. This will also be recorded and subsequently assessed.

An assistant present during the block will time two aspects of the procedure:

1. Time from first skin contact with needle to first muscle response to nerve stimulation. This will be done only on the day of surgery during the block procedure until the desired muscle twitch is elicited.
2. Time from first skin contact to completion of catheter insertion (Block time).This is done during the block procedure only on the day of surgery as noted above

Once catheter position has been assessed a total of 20 millilitres of 2% mepivacaine will be injected via the catheter in both groups. Over the subsequent 30 minutes a second blinded observer will take observations every 5 minutes to assess the degree of motor and sensory block.

The video recording of the block procedure will be sent along with the data collection form to two of the co-investigators, who will independently assess the following:

1. At the time of nerve contact by the needle, assign a rating for visibility of the needle shaft and tip according to the following scale:

   1. not visualised or poorly visualised - needle tip/shaft being isoechoic or only slightly more echogenic than background parenchyma.
   2. tip or shaft visualised with some difficulty - tip/shaft readily identified as being more echogenic than the background parenchyma but not seen in their entirety
   3. excellent visibility shaft and tip strongly echogenic relative to tissue and visualised in their entirety.
2. Assign the same rating after completion of injection
3. Judge whether circumferential and longitudinal spread of local anaesthetic is either adequate or inadequate.

Following the operation a standard infusion of 0.1% ropivacaine at 4cc/hr will be commenced via the sciatic catheter. Post operative care will be as per the standard practice at this institution.

One week post operatively the patient will be telephoned at home to check for persisting neurological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-80 years listed for total knee arthroplasty.
* ASA I-IV.
* Able to give informed consent
* Able to cooperate with study protocol.

Exclusion Criteria:

* Standard contraindication to regional anaesthesia/analgesia: local infection, coagulopathy, local anaesthetic allergy, patient refusal, diabetes mellitus, peripheral neuropathy, pre-existing nerve injury)
* Inability to consent
* Patient refusal
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Visibility of needle tip and catheter tip | Day 1
  Needle tip visibility graded by blinded observers Catheter tip visibility graded by blinded observers

SECONDARY OUTCOMES:
number of needle passes | Day 1
  The number of times the needle is withdrawn more than 2 cm and resited
success rate of block | Day 1
  Motor and sensory block will be evaluated on standard grading system every 5 minutes for 30 minutes post injection
Block procedure time | Day 1
  Time from needle insertion to the end of catheter insertion
Immediate complications | Day 1
  Vascular punctures, venous or arterial
delayed complications | One week after surgery/block
  telephone interview to elicit delayed neurologic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sugantha Ganapathy, Principal Investigator — Professor, Director, regional and Pain reseaerch
Locations (1):
- London Health Sciences Centre University Hospital, London, Ontario, Canada

REFERENCES:
- [Derived] Brookes J, Sondekoppam R, Armstrong K, Uppal V, Dhir S, Terlecki M, Ganapathy S. Comparative evaluation of the visibility and block characteristics of a stimulating needle and catheter vs an echogenic needle and catheter for sciatic nerve block with a low-frequency ultrasound probe. Br J Anaesth. 2015 Dec;115(6):912-9. doi: 10.1093/bja/aev351. PMID 26582852